CLINICAL TRIAL: NCT07197255
Title: Transcriptomic Profiling of Cumulus Cells From CAPA-IVM Cycles in Women With PCOS: A Prospective Pilot Study
Brief Title: Transcriptomic Profiling of Cumulus Cells From CAPA-IVM
Status: Recruiting | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 09/25/DD-BVMD
Record Dates: First submitted 2025-09-02; First posted 2025-09-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: PCOS (Polycystic Ovary Syndrome); Cumulus Cell; Capacitation IVM; Transcriptomic Profiling
Keywords: In vitro maturation; CAPA-IVM; Cumulus cells; Transcriptomics
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cumulus cells collected from cumulus-oocyte complexes after CAPA-IVM for transcriptomic analysis (RNA-seq).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCOS Women Undergoing CAPA-IVM: Women aged 18-38 years with PCOS (Rotterdam criteria) indicated for CAPA-IVM. From each participant, 15 cumulus-oocyte complexes (COCs) are allocated to single-culture CAPA-IVM. Cumulus cells from these COCs are collected at oocyte denudation for RNA sequencing and transcriptomic analysis.

SUMMARY:
Capacitation in vitro maturation (CAPA-IVM) has improved oocyte maturation and resulted in live births. Because cumulus cells (CCs) communicate bidirectionally with the oocyte, their transcriptomic profile may serve as a non-invasive biomarker of oocyte and embryo competence. This prospective pilot study will analyze CCs gene expression after CAPA-IVM using RNA sequencing and pathway analysis, and correlate findings with embryological outcomes including fertilization, day-3 cleavage, and blastocyst formation. Results are expected to provide insights into the molecular basis of oocyte competence and support development of non-invasive embryo selection strategies.

DETAILED DESCRIPTION:
In vitro maturation (IVM) is an alternative to conventional ovarian stimulation, particularly for women with polycystic ovary syndrome (PCOS) or at risk of ovarian hyperstimulation syndrome (OHSS). A novel technique, known as capacitation IVM (CAPA-IVM), introduces a pre-maturation step that improves both nuclear and cytoplasmic maturation and has been associated with live births. Cumulus-oocyte complexes (COCs) represent the functional unit of oocyte competence, with cumulus cells (CCs) providing bidirectional signaling that regulates oocyte development. Because CCs are routinely removed during ICSI, they serve as a readily accessible and non-invasive source of information about oocyte and embryo potential.

This prospective observational cohort study will be conducted at the IVFMD, My Duc Hospital, Ho Chi Minh City, Vietnam. Eligible participants are women diagnosed with PCOS according to the Rotterdam 2003 criteria, with serum AMH ≥ 4 ng/mL and antral follicle count (AFC) ≥ 24, indicated for CAPA-IVM treatment. From each participant, 15 COCs will be allocated to single-culture CAPA-IVM condition. CCs from each COC will be collected for transcriptomic analysis, while the oocytes are assessed for embryological outcomes. The remaining COCs will follow the standard CAPA-IVM protocol at the center.

RNA sequencing will be performed using low-input protocols. Data will undergo differential expression analysis (DESeq2), and functional interpretation using Gene Ontology and Ingenuity Pathway Analysis. Laboratory outcomes including day-3 cleavage, and blastocyst formation will be correlated with CC transcriptomic profiles. This study aims to identify non-invasive biomarkers of oocyte and embryo competence, supporting future embryo selection strategies in assisted reproduction. By correlating cumulus cell transcriptomic profiles with oocyte and embryo outcomes, this study seeks to establish preliminary non-invasive biomarkers for embryo selection in assisted reproduction.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-38 years
* BMI =< 32kg/m2
* Diagnosed with polycystic ovary syndrome (PCOS) according to the Rotterdam 2003 criteria, meet at least 2 of the following 3 features: (1) Oligo-ovulation or anovulation. (2) Clinical and/or biochemical signs of hyperandrogenism (3) Polycystic ovarian morphology on ultrasound.
* Indicated for CAPA-IVM treatment.
* Serum AMH ≥ 4 ng/mL (28.57 pmol/L).
* Antral follicle count (AFC) ≥ 24 follicles in both ovaries at the time of CAPA-IVM indication.
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Retrieved sperm from surgical procedures
* Previous IVF cycle with total immature oocytes

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with PCOS diagnosed according to the Rotterdam 2003 criteria who are indicated for CAPA-IVM treatment at IVFMD, My Duc Hospital, Ho Chi Minh City, Vietnam.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of cumulus cell transcriptomic profiles with embryological outcomes | Through study completion, an average of 1 year
  Association between cumulus cell gene expression (RNA-seq-based transcriptomic profiles) and embryological outcomes, including cleavage and embryo quality (Day 3), and blastocyst formation and grading (Days 5-6).

SECONDARY OUTCOMES:
CCs transcriptomic profiles | Through study completion, an average of 1 year
  RNA sequencing of CCs collected from individual COCs after CAPA-IVM. Differential gene expression will be analyzed using DESeq2, followed by Gene Ontology enrichment and Ingenuity Pathway Analysis to identify pathways, molecular functions, and regulatory networks associated with oocyte competence.
Number of matured oocyte | At day 2 after the Oocyte Pick-Up day
  The number of oocytes that have first polar body after denudation
Number of normal fertilized oocytes | 16-18 hours after intracytoplasmic sperm injection
  Oocytes that show the presence of two pronuclei
Number of day-3 embryos | 68 ±1 hours after intra-cytoplasmic sperm injection
  Day-3 embryo morphology assessed according to the Istanbul Consensus (2011), with reference to the revised criteria (2024)
Number of good-quality day-3 embryos | 68±1 hours after intra-cytoplasmic sperm injection
  Day-3 embryo morphology assessed according to the Istanbul Consensus (2011), with reference to the revised criteria (2024)
Number of blastocyst | Day 5 (116 ± 2 hours) and Day 6 (140 ± 2 hours) after intra-cytoplasmic sperm injection
  Blastocyst quality assessed on Day 5/6 according to the Istanbul Consensus (2011), with reference to the revised criteria (2024).
Number of good-quality blastocyst | Day 5 (116 ± 2 hours) and Day 6 (140 ± 2 hours) after intracytoplasmic sperm injection
  Good-quality blastocysts defined and graded according to the Istanbul Consensus (2011), with reference to the revised criteria (2024).
Number of frozen embryos | At the time of embryo cryopreservation
  Embryos that meet morphology and developmental criteria for cryopreservation by vitrification

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vương, PhD, MD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Background] Working Group on the update of the ESHRE/ALPHA Istanbul Consensus; Coticchio G, Ahlstrom A, Arroyo G, Balaban B, Campbell A, De Los Santos MJ, Ebner T, Gardner DK, Kovacic B, Lundin K, Magli MC, Mcheik S, Morbeck DE, Rienzi L, Sfontouris I, Vermeulen N, Alikani M. The Istanbul consensus update: a revised ESHRE/ALPHA consensus on oocyte and embryo static and dynamic morphological assessmentdagger,double dagger. Hum Reprod. 2025 Jun 1;40(6):989-1035. doi: 10.1093/humrep/deaf021. PMID 40288770
- [Background] Russell DL, Gilchrist RB, Brown HM, Thompson JG. Bidirectional communication between cumulus cells and the oocyte: Old hands and new players? Theriogenology. 2016 Jul 1;86(1):62-8. doi: 10.1016/j.theriogenology.2016.04.019. Epub 2016 Apr 21. PMID 27160446
- [Background] Assou S, Haouzi D, Mahmoud K, Aouacheria A, Guillemin Y, Pantesco V, Reme T, Dechaud H, De Vos J, Hamamah S. A non-invasive test for assessing embryo potential by gene expression profiles of human cumulus cells: a proof of concept study. Mol Hum Reprod. 2008 Dec;14(12):711-9. doi: 10.1093/molehr/gan067. Epub 2008 Nov 21. PMID 19028806
- [Background] Gebhardt KM, Feil DK, Dunning KR, Lane M, Russell DL. Human cumulus cell gene expression as a biomarker of pregnancy outcome after single embryo transfer. Fertil Steril. 2011 Jul;96(1):47-52.e2. doi: 10.1016/j.fertnstert.2011.04.033. Epub 2011 May 14. PMID 21575950
- [Background] Pham HH, Le AH, Nguyen TC, Ma MPQ, Akin N, Pham TD, Nguyen MHN, Le HL, Huynh BG, Smitz J, Ho TM, Vuong LN. Effect of single versus grouped culture of human cumulus-oocyte complexes in PCOS women treated with biphasic in vitro maturation: A sibling oocyte pilot study. Reprod Med Biol. 2024 Jun 7;23(1):e12587. doi: 10.1002/rmb2.12587. eCollection 2024 Jan-Dec. PMID 38854775
- [Background] Akin N, Richani D, Liao X, Zhao Y, Herta AC, Billooye K, Stocker WA, Mottershead DG, Harrison CA, Smitz J, Anckaert E, Gilchrist RB. Effect of cumulin and super-GDF9 in standard and biphasic mouse IVM. J Assist Reprod Genet. 2022 Jan;39(1):127-140. doi: 10.1007/s10815-021-02382-z. Epub 2022 Jan 4. PMID 34984599
- [Background] Vuong LN, Ho VNA, Ho TM, Dang VQ, Phung TH, Giang NH, Le AH, Pham TD, Wang R, Smitz J, Gilchrist RB, Norman RJ, Mol BW. In-vitro maturation of oocytes versus conventional IVF in women with infertility and a high antral follicle count: a randomized non-inferiority controlled trial. Hum Reprod. 2020 Nov 1;35(11):2537-2547. doi: 10.1093/humrep/deaa240. PMID 32974672
- [Background] Sanchez F, Lolicato F, Romero S, De Vos M, Van Ranst H, Verheyen G, Anckaert E, Smitz JEJ. An improved IVM method for cumulus-oocyte complexes from small follicles in polycystic ovary syndrome patients enhances oocyte competence and embryo yield. Hum Reprod. 2017 Oct 1;32(10):2056-2068. doi: 10.1093/humrep/dex262. PMID 28938744